CLINICAL TRIAL: NCT01896362
Title: Leishmaniasis: the Healthcare Professionals' Knowledge in Endemic Area
Brief Title: The Healthcare Professionals and the Leishmaniasis
Status: Completed | Type: Observational
Sponsor: Centro de Pesquisas René Rachou (Other Government)
Responsible Party: Principal Investigator, Carina Margonari de Souza, Carina Margonari de Souza, Centro de Pesquisas René Rachou
Other Study IDs: CentroPRR-001
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Knowledge on Leishmaniasis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this work was to investigate the healthcare professionals' knowledge about leishmaniasis in Divinópolis, an endemic county of Minas Gerais state, Brazil.

ELIGIBILITY:
Inclusion Criteria:

* work in the healthcare centers, in the case of primary care professionals;
* have a university degree for nurses, physicians, dentists and veterinarians;
* be working effectively at the time of the interview;
* accept the terms of the research through written informed consent.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nurses, physicians and dentists working in primary care units of the municipality, community health workers and zoonoses agents tied to health surveillance and veterinarians working in private veterinary clinics of Divinópolis city, Minas Gerais state, Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2010-05; Primary Completion 2010-10 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Number of questions correctly answered | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Carina M de Souza, PhD, Principal Investigator — Centro de Pesquisas René Rachou